CLINICAL TRIAL: NCT06347900
Title: Corneal Topographic Changes in Different Grades of Obstructive Sleep Apnea Syndrome
Brief Title: Corneal Topographic Changes in Different Grades of OSA
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Elshimaa A.Mateen, Clinical professor, Sohag University
Other Study IDs: Soh-Med-23-09-7PD
Record Dates: First submitted 2024-03-27; First posted 2024-04-04 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Corneal Ectasia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control group (Group1): Normal control subjects
  Interventions: Diagnostic Test: Pentacam (corneal topographic changes detection), Polysymnography
- Mild OSA (Group 2): Cases with mild obstructive sleep apnea (RDI) with respiratory distress index 5-15
  Interventions: Diagnostic Test: Pentacam (corneal topographic changes detection), Polysymnography
- Moderate OSA (Group 3): Cases with mild obstructive sleep apnea (RDI) with respiratory distress index 15-30
  Interventions: Diagnostic Test: Pentacam (corneal topographic changes detection), Polysymnography
- Sever OSA (Group4): Cases with mild obstructive sleep apnea (RDI) with respiratory distress index >30
  Interventions: Diagnostic Test: Pentacam (corneal topographic changes detection), Polysymnography

INTERVENTIONS:
Diagnostic Test: Pentacam (corneal topographic changes detection), Polysymnography — Pentacam for recording corneal parameters in different stages of OSA patients. Polysymnography for for detction of hyponea, oxygen saturation and desaturation and staging of OSA in different patients.

SUMMARY:
Corneal topographic parameters in different degrees of obstructive sleep apnea

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) syndrome is a disease characterized by recurrent total or partial upper airway collapse during sleep, interrupting or reducing the airflow, and after ward resulting in temporary awakening which causes restoration of flow of the upper airway. These intermittent complete (apnea) or partial (hypopnea) respiratory cessations decrease blood oxygen levels (hypoxia).

Upper airway stenosis causes hypoxemia and hypercapnia, which can lead to multiple organ dysfunction and is associated with systemic diseases, such as hypertension, diabetes, and coronary arteriosclerosis, and changes in the eyes include floppy eyelid syndrome, keratoconus, and glaucoma.

The prevalence of OSA is between 2% and 10% in females and 4-20% in males and obesity is a major risk factor for the development of OSA.

With all the adverse effects associated with OSA, its secondary effects cause several ocular complications. Previous studies have shown that OSA is associated with increased risks of several vision-threatening and nonthreatening ocular disorders, including senile cataracts, normal-tension glaucoma, retinal ischemia, conjunctival hyperemia, and dry eye.

Several contributory mechanisms to the ocular complications of OSA have been reported, including intermittent hypoxia, oxidative stress, systemic inflammatory responses (such as interleukin-6 (IL-6), IL-8, tumor necrosis factor-alpha (TNF-α), C-Reactive protein (CRP), matrix metalloproteinase 9 (MMP-9), vascular cell adhesion molecule (VCAM), intercellular adhesion molecule (ICAM), selectins), sympathetic system overaction, damage effects of endothelin-1, and disruption of the blood-retinal barrier (BRB) (6-8). There are limited publications that manipulate the corneal topographic parameters in different degrees of OSA, especially in the Egyptian population.

ELIGIBILITY:
Inclusion Criteria:

* patients with diagnosed OSA

Exclusion Criteria:

* Any corneal scars, previous ocular surgeries, patients with keratoconus

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: patients above age of 20 with obstructive sleep apnea syndrome with no history of previous ocular surgeries
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Keratometric readings in diopters, corneal thickness in um, average progression index value, anterior and posterior corneal elevation values. | 3 monthes
  Keratometric readings in diopters, corneal thickness in um, average progression index value, anterior and posterior corneal elevation values.

CONTACTS AND LOCATIONS:
Overall Officials: Elshimaa A.Mateen, Principal Investigator — Assistant professor of ophthalmology, Sohag University
Locations (1):
- Ophthalmology department, Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided